CLINICAL TRIAL: NCT01847079
Title: Procalcitonin to Guide Obtaining Bloodcultures in the ICU. Intensive Care Infection Score.
Brief Title: Procalcitonin to Guide Obtaining Bloodcultures in the ICU Intensive Care Infection Score
Acronym: ProBIC/ICIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, P.J. van der Geest, MD, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NL 38603.078.11
Record Dates: First submitted 2013-04-24; First posted 2013-05-06 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Procalcitonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group, procalcitonin (Other): procalcitonin to guid obtaining bloodcultures in the ICU
  Interventions: Other: Procalcitonin
- Control group, ICIS, procalcitonin (No Intervention): Measurement of PCT and ICIS.

INTERVENTIONS:
Other: Procalcitonin — Procalcitonin to guide obtaining bloodcultures
  Arms: Intervention group, procalcitonin

SUMMARY:
PROBIC

Rationale: Procalcitonin measurements can reduce the number of blood cultures in the ICU.

Objective: The investigators suggest that PCT is a marker for blood stream infection in all patients in the ICU in whom attending physicians/ intensivists order blood culturing in the suspicion of microbial infection. The investigators want to demonstrate that its use for guiding blood culturing is cost-effective and safe compared with blood cultures alone.

Study design: Prospective, non- inferiority, multicenter, single-blinded, cluster- randomised cross-over clinical trial.

Intervention (if applicable): The intensive care units will be allocated into two groups: a control group (blood culture) and the intervention group (procalcitonin).

Main study parameters/endpoints: Safety, expressed as mortality at day 28 and 90, with a mortality difference not exceeding a between groups difference of 10% by non-inferiority analysis.

Cost-effectiveness, expressed in euro, calculated by deducting costs of procalcitonin testing from saved blood cultures compared with standard treatment spending on blood cultures in the control group.

ICIS

Rationale: The aim was to evaluate the Intensive Care Infection Score (ICIS) in predicting microbial infection and its sequelae in critically ill patients in whom attending physicians/ intensivists order blood culturing in the suspicion of microbial infection.

Objective: Because of the complexity of the pathophysiology of systemic inflammation it is unlikely that a single parameter will have sufficient diagnostic accuracy for infection. Therefore we will study combining parameters producing a diagnostic score.

Study design: Prospective, multicenter, cohort trial. Supplement for the control arm of the ProBIC study.

Intervention (if applicable): Blood is drawn for daily routine laboratory measurements and collected in K3EDTA aliqnots. The ICIS score is composed of five blood-cell derived parameters which can be extracted using the same aliqnots.

Main study parameters/endpoints: To develop and evaluate a blood- cell derived score to enable the diagnosis of microbial infection, its likelihood, its invasiveness and severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients will need to be over the age of 18 and suffering from an assumed infection deemed clinically worthy for blood culturing.

Exclusion Criteria:

* Uncontrolled malignancy
* Immunosuppressive or immunostimulatory therapy
* Neutropenia, defined as leukocyte count less then 0.5x109/L
* Moribund patients
* Predetermined illness with an expected death within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
1. Safety, expressed as mortality at day 28 and 90, with a mortality difference not exceeding a between groups difference of 10% by non-inferiority analysis. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick van der Geest, MD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland

REFERENCES:
- [Derived] van der Geest PJ, Mohseni M, Nieboer D, Duran S, Groeneveld ABJ. Procalcitonin to guide taking blood cultures in the intensive care unit; a cluster-randomized controlled trial. Clin Microbiol Infect. 2017 Feb;23(2):86-91. doi: 10.1016/j.cmi.2016.10.004. Epub 2016 Oct 13. PMID 27746396
- [Derived] van der Geest PJ, Mohseni M, Linssen J, Duran S, de Jonge R, Groeneveld AB. The intensive care infection score - a novel marker for the prediction of infection and its severity. Crit Care. 2016 Jul 7;20(1):180. doi: 10.1186/s13054-016-1366-6. PMID 27384242